CLINICAL TRIAL: NCT00002125
Title: A Multicenter Study of Oral Versus Intravenous Hydration in AIDS Patients With CMV Retinitis Treated With Foscavir (Foscarnet Sodium)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astra USA (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 020H; 93-FOS-31
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-06

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Infusions, Intravenous; Foscarnet; Cytomegalovirus Infections; Administration, Oral; Acquired Immunodeficiency Syndrome; Fluid Therapy
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet

INTERVENTIONS:
Drug: Foscarnet sodium

SUMMARY:
To assess the relative efficacy of oral versus intravenous hydration during foscarnet sodium (Foscavir) induction therapy, as determined by changes in creatinine clearance. To estimate the timing and volume of oral fluid hydration required to establish a diuresis before and during intravenous Foscavir therapy. To assess the general tolerance of two hydration regimens by the adverse event profile associated with each.

DETAILED DESCRIPTION:
Patients are randomized to receive oral hydration versus intravenous hydration therapy during concomitant intermittent intravenous Foscavir therapy for treatment of cytomegalovirus (CMV) retinitis. Treatment continues during 2 or 3 weeks of induction Foscavir therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* Recent diagnosis of CMV retinitis, by ophthalmoscopic appearance, that requires induction therapy.
* No corneal, lens, or vitreous opacification that precludes examination of the fundi.
* No evidence of other end organ CMV infection.
* No evidence of tuberculous, diabetic, or hypertensive retinopathy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Clinically significant cardiac, pulmonary, neurologic, gastrointestinal or renal impairment that would prevent adequate voluntary oral hydration (e.g., intubation, coma, status post-gastrectomy, colon resection, gastrointestinal tumors, malabsorption, chronic diarrhea) OR with which hydration would be hazardous (e.g., congestive heart failure).
* Known allergy to foscarnet or related compounds.
* Considered noncompliant or unreliable for study participation.

Concurrent Medication:

Excluded:

* Any investigational drug.
* Potentially nephrotoxic drugs (e.g., amphotericin B, aminoglycosides, cisplatin).

Prior Medication:

Excluded:

* Any investigational drug within 28 days prior to study entry.
* Potentially nephrotoxic drugs (e.g., amphotericin B, aminoglycosides, cisplatin) within 7 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112

CONTACTS AND LOCATIONS:
Overall Officials: Wool GM, Study Chair
Locations (11):
- United States (11):
  - Dr Ralph Hansen, Beverly Hills, California
  - Dr Milan Fiala, Los Angeles, California
  - Dr G Michael Wool, Los Angeles, California
  - AIDS Community Research Consortium, Redwood City, California
  - Ingenix Kern McNeill Decatur, Atlanta, Georgia
  - Dr John Karedes, Indianapolis, Indiana
  - Dr Paul Benson, Berkley, Michigan
  - Dr Ronald Nahass, Somerville, New Jersey
  - Dr Ronald J Grossman, New York, New York
  - Community Health Network, Rochester, New York
  - Austin Infectious Disease Consultants, Austin, Texas